CLINICAL TRIAL: NCT05467215
Title: Can Brief Exposure to Hyperoxia Improve Function After Chronic Spinal Cord Injury?
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Pro00061817
Record Dates: First submitted 2022-07-06; First posted 2022-07-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
Keywords: Hypoxia; Hyperoxia; Reflex; Sensation
MeSH Terms: conditions — Spinal Cord Injuries; Hypoxia; Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized crossover design
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants with SCI will be masked. The experimenter collecting the sensory data and the experimenter analyzing the reflex data will be masked to the oxygen/air exposure, to avoid bias. The participant and the experimenter will be unmasked once all data collection has been completed for the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyperoxia followed by room air (Experimental): Group 1 will receive oxygen (99%) in Phase 1, and room air (placebo) in Phase 2. Each phase will consist of 2 experiments. In Phase 1, the first experiment will test skin sensation using von Frey Hairs, while the second experiment will test a cutaneous reflex. In Phase 2, the first experiment will test the cutaneous reflex, while the second experiment will test skin sensation with von Frey Hairs. Both high oxygen and room air will be delivered through a face mask. The flow rate will be 10 litres/min for a 2-min period. Participants and experimenters will be blinded to the intervention. Measures will be taken before and after each exposure. In this way, each participant will be involved in four experimental sessions with a minimum of 2-week intervals between every testing session. Each experimental session will take approximately 1.5 to 2 hours. A total duration of involvement in the study is a minimum of 7 weeks.
  Interventions: Drug: Pure oxygen (99%) from Praxair, Edmonton, DIN# 02014408
- Room air followed by hyperoxia (Placebo Comparator): Group 2 will receive room air (placebo) in Phase 1, and oxygen (99%) in Phase 2. Each phase will consist of 2 experiments. In Phase 1, the first experiment will test the cutaneous reflex, while the second experiment will test skin sensation with von Frey Hairs. In Phase 2, the first experiment will test skin sensation using von Frey Hairs, while the second experiment will test a cutaneous reflex. Both high oxygen and room air will be delivered through a face mask approved by Health Canada. The flow rate will be 10 litres/min for a 2-min period. Participants and experimenters will be blinded to the intervention. Measures will be taken before and after each exposure.In this way, each participant will be involved in four experimental sessions with a minimum of 2-week intervals between every testing session. Each experimental session will take approximately 1.5 to 2 hours. A total duration of involvement in the study is a minimum of 7 weeks.
  Interventions: Drug: Pure oxygen (99%) from Praxair, Edmonton, DIN# 02014408

INTERVENTIONS:
Drug: Pure oxygen (99%) from Praxair, Edmonton, DIN# 02014408 — Participants will receive oxygen (99%) or room air (placebo) delivered through a face mask at a flow rate of 10 litres/min for 2 minutes. The participants will be exposed twice to both conditions over 4 experiments at a minimum of 2 week intervals between each testing session.
  Other Names: Compressed air from Praxair, DIN# 02014483

SUMMARY:
This proof-of-principle study will determine if breathing an increased concentration of oxygen above the concentration in normal room air results in changes in the sensory and motor function in people with subacute or chronic, severe spinal cord injury (SCI).

DETAILED DESCRIPTION:
This proof-of-principle study will include a small number of participants with subacute or chronic (>3 months post-injury), severe spinal cord injury (i.e., AIS A, B or C). After screening for potential contraindications, participants will attend 4 experimental sessions. In each session, their sensory or reflex function will be tested at regular intervals. Once baseline recordings are established, participants will be given either room air or 99% oxygen to breathe through a face mask for 2 minutes. It will be determined if breathing 99% oxygen results in a change in the sensory and motor functions recorded before and shortly after breathing oxygen.

Administration of a high concentration of oxygen at atmospheric pressure for a short duration has been completed without adverse effects in healthy individuals, and individuals with various forms of injury including chronic obstructive lung disease, traumatic brain injury, stroke, and spinal cord injury. Duration of administration has ranged from 3 min to 4 hours without adverse effects.

If this initial trial indicates that improvements in sensory and motor function are induced by this short exposure, exploration of therapeutic ways to increase blood flow to the spinal cord will be undertaken

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with traumatic SCI with onset ≥3 months prior,
2. Between 18 - 65 yr old,
3. ASIA Impairment Scale at discharge classified as A, B or C,
4. Injury level between C5 and T10,
5. Able to give informed, written consent.

Exclusion Criteria:

1. Frequent uncontrolled autonomic dysreflexia,
2. Uncontrolled high blood pressure,
3. Cardiac or cardiovascular disease,
4. Cancer,
5. Active urinary tract infection,
6. Active pressure sores,
7. Signs of deep vein thrombosis in the legs,
8. Severe swelling of the feet and/or legs,
9. Severe cognitive impairment,
10. Pulmonary dysfunction such as chronic obstructive pulmonary disease or acute respiratory infection,
11. Any condition which would be exacerbated by sitting or lying in one position for 2 hours, such as low back pain
12. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin Sensation | Pre-intervention (exposure to high oxygen)
  Quantification using von Frey Hairs at three locations above and below the level of injury.
Skin Sensation | Immediately after intervention (exposure to high oxygen)
  Quantification using von Frey Hairs at three locations above and below the level of injury.
Skin Sensation | Pre-intervention (exposure to room air)
  Quantification using von Frey Hairs at three locations above and below the level of injury.
Skin Sensation | Immediately after intervention (exposure to room air)
  Quantification using von Frey Hairs at three locations above and below the level of injury.

SECONDARY OUTCOMES:
Reflex Excitability | Pre-intervention (exposure to high oxygen)
  Elicited by electrical stimulation of the skin on the arch of the foot and measured by surface electromyography (EMG).
Reflex Excitability | Immediately after intervention (exposure to high oxygen)
  Elicited by electrical stimulation of the skin on the arch of the foot and measured by surface electromyography (EMG).
Reflex Excitability | Pre-intervention (exposure to room air)
  Elicited by electrical stimulation of the skin on the arch of the foot and measured by surface electromyography (EMG).
Reflex Excitability | Immediately after intervention (exposure to room air)
  Elicited by electrical stimulation of the skin on the arch of the foot and measured by surface electromyography (EMG).

CONTACTS AND LOCATIONS:
Overall Officials: Jaynie Yang, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Clinical Sciences Bldg, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT05467215/Prot_000.pdf